CLINICAL TRIAL: NCT02007928
Title: Assessment of Incidence of Adverse Events in a Naive Pediatric Population Treated With an (Typical and Atypical) Antipsychotic Drug Over 12 Months Follow-up
Brief Title: Assessment of Adverse Events in a Naive Pediatric Population Treated With an Antipsychotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12-PP-12
Record Dates: First submitted 2013-04-23; First posted 2013-12-11 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Dissociative Disorders; Schizophrenia
MeSH Terms: conditions — Dissociative Disorders; Schizophrenia | interventions — Risperidone; Aripiprazole; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rispéridone, aripiprazole, olanzapine... (Other): Study:
  We propose a prospective, interventional multicenter study.
  Method:
  Both in and out patients may be included in the study Patients will be recruited over a period of 24 months. They will be followed up for 12 months. Each patient will receive one year of therapeutic monitoring after the introduction of the antipsychotic drug.
  The therapeutic monitoring will include clinical, electrocardiographical, and laboratory assessments. These assessments are performed at baseline (before prescribing treatment) and at 1 month (M1), at 3 months (M3), 6 months (M6), 9 months (M9), and at 12 months (M12) after the first prescription of the antipsychotic drug.
  Interventions: Other: Rispéridone, aripiprazole, olanzapine

INTERVENTIONS:
Other: Rispéridone, aripiprazole, olanzapine — Study:
  We propose a prospective, interventional multicenter study.
  Method:
  Both in and out patients may be included in the study Patients will be recruited over a period of 24 months. They will be followed up for 12 months. Each patient will receive one year of therapeutic monitoring after the introduction of the antipsychotic drug.
  The therapeutic monitoring will include clinical, electrocardiographical, and laboratory assessments. These assessments are performed at baseline (before prescribing treatment) and at 1 month (M1), at 3 months (M3), 6 months (M6), 9 months (M9), and at 12 months (M12) after the first prescription of the antipsychotic drug.

SUMMARY:
We propose a prospective multicenter study, whose originality lies in the inclusion of the naive child and adolescent population. Its purpose is to evaluate the incidence of adverse events related to the use of l antipsychotic drugs in children and adolescents with no history of taking such drugs.

The inclusion criteria will be: (1) male or female inpatients, (2) aged from 6 to 18 years, (3) requiring antipsychotic treatment, (4) receiving antipsychotic drug for less than 28 days without taking antipsychotic before or with a history of antipsychotic over a maximum period of three consecutive months and discontinued for at least 6 months.

Therapeutic monitoring during the 12 month study period will include clinical assessments and laboratory testing. These assessments will be performed before treatment (at inclusion), and at 1, 3, 6, 9, 12 months after the introduction of the antipsychotic drug.

DETAILED DESCRIPTION:
a prospective multicenter study, whose originality lies in the inclusion of the naive child and adolescent population

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Aged from 6 to 18 years
* In whom antipsychotic treatment is indicated
* Who have never been treated with antipsychotic medication (other than metoclopramide (Primperan®) for pediatric indications) or with a history of antipsychotic over a maximum period of three consecutive months and discontinued for at least 6 months. .

The non-inclusion criteria:

* Any

The exclusion criteria:

* Refusal or withdrawal of consent by the patient or his/her parents.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Clinical assessment and laboratory | 12 months
  1. Clinical Assessment A: General assessment of adverse events by the Pediatric Adverse Event Rating Scale (PAERS-Clinician) (March et al, 2007). Performed at each visit.
     B: Somatic parameters to be monitored: weight, size, body mass index (BMI), abdominal perimeter, blood pressure, temperature. Performed at each visit.
     C: Electrocardiographic assessment of QT interval D: Neuromuscular adverse events: Abnormal Involuntary Movement Scale (AIMS) (Guy, 1976a), Barnes Akathisia Rating Scale (BARS) (Barnes, 1989), Simpson Angus Scale (SAS) (Simpson and Angus, 1970), Bush Francis Catatonia Rating Scale (BFCRS) (Bush and al, 1996),
  2. Laboratory assessments. The following laboratory tests will be obtained on each visit: complete blood count, liver enzymes, creatine phosphokinase, glycemia, cholesterol (total, light, and heavy), triglycerides, CRPus, prolactin, insulin, HOMA, HbA1C, vitamin D.

SECONDARY OUTCOMES:
Risk Factors | 12 months
  Tanner score of puberty at inclusion: population will be divided into three groups: prepubertal (stage ≤ 1); currently in puberty (stages 2 to 4) and puberty adult (stage 5).
  Drug history: age at initiation of treatment, the first-line atypical antipsychotic drug, other treatment(s), age of onset of disorder for which the prescription of an atypical antipsychotic drug was indicated.
  The diagnosis is made using the Schedule for Affective Disorders and Schizophrenia for School Age Children (Kiddie-SADS) (Kaufman and al, 1997).
Persistence and/or reversibility of adverse events before the end of the study | 12 months
  The investigators propose the following definitions for this study, based on published data and our preliminary study:
  * A persistent adverse event is an event that is still present 3 months after treatment cessation
  * A reversible adverse event is an event that has fully resolved 3 months after treatment cessation
Scores | 12 months
  4) Evaluation of the evolution of disorder severity at baseline, at M1, M3, M6, M9 and M12 The clinical severity of the disorder will be assessed using the Clinical Global Impressions Scales (CGI) (Guy, 1976b).
  5) Evaluation of the evolution of social functioning at baseline, at M6 and at M12 Social functioning will be assessed by the Child Global Assessment Scale (CGAS).
  6) Evaluation of the evolution of therapeutic alliance at M1, at M3, M6, M9 and at M12
Quality of life | 12 months
  7) Evaluation of the evolution of quality of life at baseline, at M1, M3, M6, M9 and at M12 Quality of life will be assessed by the Sheehan Disability Scale 8) The evaluation of the evolution of eating disorder at baseline, at M1, M3, M6, M9 and at M12 will be assessed by the Questionnaire of Eating and Weight Patterns 9) The evaluation of the evolution of physical activity at baseline, at M1, M3, M6, M9 and at M12 will be assessed by Dennison measure 10) Evaluation of the evolution of DSM diagnosis at baseline and at M12 by the Schedule for Affective Disorders and Schizophrenia for School Age Children (Kiddie-SADS)

CONTACTS AND LOCATIONS:
Overall Officials: MENARD Marie-Line, PH, Study Chair — CHU de Nice - 52 avenue de la Californie 06 200 Nice
Locations (14):
- France (14):
  - CH de Cannes, Cannes, Alpes-maritimes
  - Service de psychiatrie de l'enfant et de l'adolescent, Nice, Alpes-Maritimes
  - CH D'antibes, Antibes, Alpes-Maritime
  - CH Henri laborit, Poitiers, Charente Maritime
  - Fondation Vallée, Gentilly, Paris
  - Ch le Vinatier, Bron
  - CHRU de Lille, Lille
  - Centre Hospitalier Spécialisé Esquirol, Limoges
  - CH St Jean de Dieu, Lyon
  - HCL, Lyon
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - AP-HP, Paris
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Menard ML, Thummler S, Giannitelli M, Olliac B, Bonnot O, Cohen D, Askenazy F; ETAPE Study group. Incidence of adverse events in antipsychotic-naive children and adolescents treated with antipsychotic drugs: a French multicentre naturalistic study protocol (ETAPE). BMJ Open. 2016 Apr 6;6(4):e011020. doi: 10.1136/bmjopen-2015-011020. PMID 27053275